CLINICAL TRIAL: NCT02782208
Title: Lipolytic Effects of GH in Hypopituitary Patients in Vivo: Molecular Mechanisms and Temporal Patterns.
Brief Title: Lipolytic Effects of GH in Hypopituitary Patients in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: GHD01
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2017-10

CONDITIONS: Hypopituitarism; Insulin Resistance; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Pituitary Diseases; Brain Diseases
MeSH Terms: conditions — Hypopituitarism; Insulin Resistance; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Pituitary Diseases; Brain Diseases | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acipimox/GH substitution (Active Comparator): Drug: Acipimox Tablet Acipimox 250 mg administered 4 times previous to and during the investigation day Other Name: Tablet Olbetam 250 mg Continue GH substitution as usually.
  Interventions: Drug: Acipimox; Drug: GH substitution
- Acipimox/GH pause (Active Comparator): Drug: Acipimox Tablet Acipimox 250 mg administered 4 times previous to and during the investigation day Other Name: Tablet Olbetam 250 mg Pause GH substitution to days prior to the study day.
  Interventions: Drug: Acipimox; Other: GH pause
- Placebo/GH substitution (Placebo Comparator): Drug: Placebo tablets Continue GH substitution as usually.
  Interventions: Drug: Placebo; Drug: GH substitution
- Placebo/GH pause (Placebo Comparator): Drug: Placebo tablets Pause GH substitution to days prior to the study day.
  Interventions: Drug: Placebo; Other: GH pause

INTERVENTIONS:
Drug: Acipimox — Acipimox is administered 4 times previous to and during the investigation day. Acipimox is used to suppress the lipolytic effect of GH.
  Other Names: Olbetam
  Arms: Acipimox/GH pause; Acipimox/GH substitution
Drug: Placebo — Placebo is administered 4 times previous to and during the investigation day.
  Arms: Placebo/GH pause; Placebo/GH substitution
Drug: GH substitution — GH substitution as usually
  Arms: Acipimox/GH substitution; Placebo/GH substitution
Other: GH pause — GH substitution pause two days prior to the experimental day
  Arms: Acipimox/GH pause; Placebo/GH pause

SUMMARY:
Growth hormone (GH) is essential for longitudinal bone growth and somatic development. These protein anabolic effects require sufficient nutritional supply. During fasting and caloric restriction GH predominantly promotes fat metabolism.

GH counteracts the effect of insulin in many tissues, of which insulin-stimulated glucose uptake in skeletal muscle has been most extensively studied. Substrate competition between elevated free fatty acids and glucose is suggested as a mechanism, and this hypothesis can be tested mechanistically by means of acipimox, which is a nicotinic acid that suppresses the fat metabolizing effects of GH.

The hypothesis is, that the suppressive effect of GH on insulin-stimulated glucose uptake in skeletal muscle is obviated by acipimox-induced inhibition of fat metabolism.

In order to investigate this, eight adult hypopituitary patients with documented GH-deficiency will be studied in the presence and absence of GH and acipimox, respectively, and biopsies from skeletal muscle and subcutaneous adipose tissue will be analyzed.

Knowledge of the effects of growth hormone and fat metabolism can in shot-sight as well as in long-sight have great importance for the understanding of growth disorders from overweight and type 2 diabetes to malnutrition and eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* hypopituitary patients with documented GH-deficiency

Exclusion Criteria:

* other significant disease

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Lipolytic activity measured as area under the curve (AUC) for FFA (free fatty acid) before and during clamp-conditions. | 1 year

SECONDARY OUTCOMES:
GH signaling proteins and gene targets in adipose and skeletal muscle tissues measured by western blotting and qPCR | 1,5 years
Insulin sensitivity as measured by M value and GIR (glucose infusion rate) | 6 months
Substrate metabolism as measured by indirect calorimetry, tritiated glucose and circulating hormones and metabolites | 1 year
PDH (pyruvate dehydrogenase) activity in skeletal muscle measured by an PDH activity assay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Principal Investigator — University Hospital of Aarhus
Locations (1):
- University Hospital of Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tunaru S, Kero J, Schaub A, Wufka C, Blaukat A, Pfeffer K, Offermanns S. PUMA-G and HM74 are receptors for nicotinic acid and mediate its anti-lipolytic effect. Nat Med. 2003 Mar;9(3):352-5. doi: 10.1038/nm824. Epub 2003 Feb 3. PMID 12563315
- [Background] Nellemann B, Vendelbo MH, Nielsen TS, Bak AM, Hogild M, Pedersen SB, Bienso RS, Pilegaard H, Moller N, Jessen N, Jorgensen JO. Growth hormone-induced insulin resistance in human subjects involves reduced pyruvate dehydrogenase activity. Acta Physiol (Oxf). 2014 Feb;210(2):392-402. doi: 10.1111/apha.12183. Epub 2013 Nov 22. PMID 24148194
- [Background] Clasen BF, Poulsen MM, Escande C, Pedersen SB, Moller N, Chini EN, Jessen N, Jorgensen JO. Growth hormone signaling in muscle and adipose tissue of obese human subjects: associations with measures of body composition and interaction with resveratrol treatment. J Clin Endocrinol Metab. 2014 Dec;99(12):E2565-73. doi: 10.1210/jc.2014-2215. PMID 25050904
- [Background] Krusenstjerna-Hafstrom T, Clasen BF, Moller N, Jessen N, Pedersen SB, Christiansen JS, Jorgensen JO. Growth hormone (GH)-induced insulin resistance is rapidly reversible: an experimental study in GH-deficient adults. J Clin Endocrinol Metab. 2011 Aug;96(8):2548-57. doi: 10.1210/jc.2011-0273. Epub 2011 May 25. PMID 21613350
- [Background] Nielsen TS, Jessen N, Jorgensen JO, Moller N, Lund S. Dissecting adipose tissue lipolysis: molecular regulation and implications for metabolic disease. J Mol Endocrinol. 2014 Jun;52(3):R199-222. doi: 10.1530/JME-13-0277. Epub 2014 Feb 27. PMID 24577718
- [Background] Moller N, Jorgensen JO. Effects of growth hormone on glucose, lipid, and protein metabolism in human subjects. Endocr Rev. 2009 Apr;30(2):152-77. doi: 10.1210/er.2008-0027. Epub 2009 Feb 24. PMID 19240267
- [Background] Nielsen S, Moller N, Christiansen JS, Jorgensen JO. Pharmacological antilipolysis restores insulin sensitivity during growth hormone exposure. Diabetes. 2001 Oct;50(10):2301-8. doi: 10.2337/diabetes.50.10.2301. PMID 11574412
- [Derived] Hjelholt AJ, Charidemou E, Griffin JL, Pedersen SB, Gudiksen A, Pilegaard H, Jessen N, Moller N, Jorgensen JOL. Insulin resistance induced by growth hormone is linked to lipolysis and associated with suppressed pyruvate dehydrogenase activity in skeletal muscle: a 2 x 2 factorial, randomised, crossover study in human individuals. Diabetologia. 2020 Dec;63(12):2641-2653. doi: 10.1007/s00125-020-05262-w. Epub 2020 Sep 18. PMID 32945898